CLINICAL TRIAL: NCT03171571
Title: Personal Lifestyle Assistant for Better Health Through Nutrition : Cook to Health Study
Brief Title: Personal Lifestyle Assistant for Better Health Through Nutrition
Acronym: C2H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Université Joseph Fourier (Other); AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC16.019
Record Dates: First submitted 2017-04-11; First posted 2017-05-31 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: eating Behavior; Volunteers
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Coaching procedure (Experimental): Volunteers will received Updated National Dietary Guidelines about food and physical activity with a one year follow-up, plus connected coaching.
  Interventions: Other: Coaching procedure

INTERVENTIONS:
Other: Coaching procedure — In this study, the volunteers will be followed during one year. The wellbeing will be followed with :
  * survey like FFQ, SF36, dietary habits.
  * actimetry measurement
  * one year follow-up of weight, waist measurement
  * nutritional biomarkers

SUMMARY:
Unhealthy lifestyles are major factors contributing to chronic conditions that impose a huge financial burden in EU healthcare systems. Unfortunately, the communication of Public Health failed to influence consumer to change their habits. In this study, the aim is to evaluate the impact of a regular monitoring during 1 year on wellbeing and dietary habits in healthy volunteers.

DETAILED DESCRIPTION:
Today, medicine mainly curative and reactive is primarily interested in sick people. Now, with our aging Western populations, we face a strong increase in chronic diseases incidence / prevalence that have a financial cost that becomes unbearable. Society's resources are being drained by the rising costs of disease management and of incremental improvements to our existing health care system. Immediate action is required to reverse these trends. The paradigm shift would be to move from a reactive to a proactive medicine that promote healthy life style to decrease incidence of chronic conditions through P4 Medicine that is Preventive, Participative, Predictive and Personnalized. However, unhealthy lifestyles are major factors contributing to chronic conditions that impose a huge financial burden in EU healthcare systems. Insufficient physical activity, poor diet and obesity are significant risk factors for cancers, cardiovascular, chest, metabolic disorders and leading causes of morbidity and premature mortality. Clinically studies indicate that different conditions can be prevented and sometimes reversed through adaptation of healthy habits. But the communication of Public Health failed to influence consumer to change their habits. Hence, it is recognized as a gold standard that better nutrition and better health will reduce the risk of chronic diseases such as obesity and cardiovascular diseases, which impact heavily on health spending.

A report by the French National Assembly estimated the cost of obesity for the health insurance, if we add the daily allowances of sick care costs, between 2 and 6 € billion / year (until 4.6% of current health expenditure). As recently summarized by Caroline K. Kramer I 2015 moderate weight loss is related to favorable clinical outcomes. A weight loss of 7% (modification of lifestyle) reduced diabetes progression (-58%). The data collected addressed to health professionals will also enable better guide diagnostics and more efficient care strategies. Unfortunately free-living individuals are often poor at judging the healthiness of their own diet (choice of meal constituents, cooking methods, and portion sizes pattern of eating). Moreover, there is a lack of awareness of the contextual features influencing eating behavior and even where there is motivation to change, people have difficulty translating good intentions into healthy behaviors. Hence, their day-to-day constraints (lack of time, lack of knowledge, constraining family and cultural habits, personal tastes) make it difficult for them to comply and adopt the nationally recommended healthy lifestyles. In this study, the volunteers will be followed during one year.

The wellbeing will be followed with :

* survey like FFQ, SF36, dietary habits.
* actimetry measurement
* one year follow-up of weight, waist measurement
* nutritional biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults based in Grenoble area France without known chronic medications (except contraception) or recent surgical intervention or hospitalization (< 6 months);
* Be able to understand and follow the protocol and use the personal health monitoring devices;
* Be the owner of a electronic tablet (iOS or Android platform) and have a valid Internet connection with access from home;
* Be able to understand the study, its aim and methodology
* Be legally able to give consent.
* 25 < BMI < 29
* 35 y <Age < 45 y
* Live as a couple and and be the main person who prepares meals

Exclusion Criteria:

Vital prognosis engaged within 6 months;

* Smoker
* Being unable to understand, follow objectives and methods due to cognition or language problems;
* Be under chronic use of medications;
* Be likely to move away from the geographic inclusion zone (mainland France);
* Be unavailable (e.g. work commitment abroad) for the two months following inclusion;
* Pregnant women, feeding and parturient
* Playing sports at a high level
* Subject under administrative or judicial control
* All eating disorders

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Alternate Healthy Eating Index-2010 (AHEI-2010) score | over a 1-year period
  calculated by Food Frequency Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PISON, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Universiy Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No